CLINICAL TRIAL: NCT03845218
Title: A Survey Study of Retinitis Pigmentosa (RP) Clinical Measures and Repeatability Testing of Potential Outcome Measures.
Brief Title: Retinitis Pigmentosa Clinical Measures and Repeatability Testing of Potential Outcome Measures
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190056; 19-EI-0056
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10-01

CONDITIONS: Retinitis Pigmentosa
Keywords: Retina; Imaging; Psychophysics; Functional Outcome Measures; Natural History
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Participants without RP
- Participants with RP: Participants must have evidence of RP as defined by characteristic ERG responses, visual fields, clinical exam and/or genetic testing

SUMMARY:
Background:

Retinitis pigmentosa (RP) is a group of blinding eye diseases. It is caused mostly by mutations in photoreceptor-expressed genes. RP affects about 2 million people globally. There is no cure, but treatment and diagnosis can be guided by certain tests. Researchers want to see how well these tests capture stages of RP.

Objectives:

To find out how well certain tests track changes in retinitis pigmentosa.

Eligibility:

People ages 12 and older with RP

Healthy volunteers ages 18 and older with no evidence of RP

Design:

Participants will be screened in another protocol.

Participants will have 2 visits about 6 weeks apart. Both will include all the tests below. Each visit will last 5-6 hours, or a visit can be split into 2 days.

Participants will give their medical and eye history.

Participants will have an eye exam. Their pupils will be dilated with eye drops.

Participants will give blood samples.

Pictures of participants retinas will be taken. Their retinas will be measured.

Participants will take several eye tests. They will:

Sit in a dark room and press a button when they see lights.

View a bright background then press a button when they see lights.

Look into a bowl and press a button when they see lights.

Sit in the dark with their eyes patched. Then they will take eye-numbing drops and wear contacts as lights flash. A small electrode taped to their forehead will record signals from their retinas.

Minors will give written consent to stay in the study when they turn 18. After the study ends, they may also be asked to give consent for researchers to continue to use their study information.

DETAILED DESCRIPTION:
Precis

Objective: The objective of this study is to investigate the nature of photoreceptor dysfunction in retinitis pigmentosa (RP) patients using focal static and kinetic psychophysical tests to develop functional outcome measures for the clinical trial study in RP. Correlation of novel spatial functional maps with other functional measures (such as visual acuity and multifocal electroretinography) will help provide a full description of functional change. Employing new imaging methods to visualize and analyze structural changes in the retina will allow for the evaluation of structural changes that underlie disease progression. Developing these measures has the potential to advance the field by elucidating the process of photoreceptor degeneration as well as being a scaffold for which candidate therapies could be trialed.

Study Population: Up to 120 participants with a diagnosis of RP will be enrolled. Up to

30 healthy volunteers will also be enrolled for a total accrual ceiling of 150.

Design: This is a single center, observational, cross-sectional repeatability study of patients with retinitis pigmentosa. The goal of Aim 1 is to identify measures that could be used in future studies to track the extent of functional retina over time. The goal of Aim 2 is to evaluate structural measures for RP. The goal of Aim 3 is to assess the participant s performance on questionnaires assessing visual function. The goal of Aim 4 is to survey the cytokine/lymphokine profile.

Outcome Measures: The primary outcome measure will be the limits of agreement in repeatability calculations of the tests performed. Secondary outcome measures will include analysis of parameter testing based on severity groups. Macular thickness as measured by optical coherence tomography (OCT), as well as ellipsoid zone band length will be quantified. Functional testing with photopic perimetry and scoptopic perimetry and kinetics will be quantified. Multifocal electroretinography (mfERG) will be analyzed by subfield and possible ring analyses. Correlations of questionnaire scores with objective measures will be analyzed.

ELIGIBILITY:
* INCLUSION CRITERIA for RP Participants:

To be eligible, the following inclusion criteria must be met, where applicable.

* Participant must be 12 years of age or older.
* Participant (or legal guardian) must understand and sign the protocol s informed consent document.
* Participant must have evidence of RP as defined by characteristic ERG responses, visual fields, clinical exam and /or genetic testing.

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

To be eligible, the following inclusion criteria must be met:

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol s informed consent document.
3. Participant must not have evidence of RP.

EXCLUSION CRITERIA FOR ALL PARTICIPANTS:

A participant is not eligible if any of the following exclusion criteria are present.

* Participant is actively receiving study therapy in another investigational study.
* Participant is started on (or changed dosage of) topical or systemic carbonic anhydrase inhibitor (CAI) treatment in the three months prior to enrollment.
* Participant is expected to be unable to comply with study procedures or follow-up visits.
* Participant has evidence of an ocular disease other than RP in either eye that may confound the outcome of the study (e.g., diabetic retinopathy with ten or more hemorrhages or microaneurysms, uveitis, pseudovitelliform macular degeneration, severe myopia).
* Participant is taking ocular or systemic medications known to be toxic to the lens, retina or optic nerve (e.g., ethambutol, chloroquine, or hydroxychloroquine).
* Participant has a condition that would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control) by interfering with the participant s ability to engage in the required protocol evaluation and testing and/or comply with study visits.
* Participant is an NIH employee associated with this study.
* Participant is unable or unwilling to give informed consent that includes use of medical records and clinical samples for current and future research.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 120 participants aged 12 or older with a diagnosis of RP. Up to 30 healthy volunteers.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Macular thickness as measured by OCT, EZ band length; functional testing including photopic/scotopic perimetry and kinetics, mfERG | ongoing
  The primary outcome measure will be the limits of agreement in repeatability calculations of the tests performed.

SECONDARY OUTCOMES:
Secondary outcome measures will include analysis of parameter testing based on absolute measures to categorize testing results into severity groups | ongoing
  Information about which tests did not yield quantifiable measures in which participants will also be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Laryssa A Huryn, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-EI-0056.html